CLINICAL TRIAL: NCT06189638
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy and Safety of Antimicrobial Peptide PL-5 Topical Spray in Patients With Mild Infections of Diabetic Foot Ulcers
Brief Title: Phase II Study to Evaluate Efficacy and Safety of AMP Peptide PL-5 in Mild Infections of Diabetic Foot Ulcers
Acronym: PL-5
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu ProteLight Pharmaceutical & Biotechnology Co., Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 280800-JSPL-PL-5-203
Record Dates: First submitted 2023-12-06; First posted 2024-01-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetic Foot Infection; Diabetic Foot; Diabetic; Wound Infection
MeSH Terms: conditions — Diabetic Foot; Wound Infection

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized (1:1:1) to receive twice a day, 14 days treatment of Antimicrobial Peptide PL-5 Topical Spray (1‰), Antimicrobial Peptide PL-5 Topical Spray (2‰) and placebo of Antimicrobial Peptide PL-5 Topical Spray (vehicle).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Antimicrobial Peptide PL-5 Topical Spray and placebo will not be identical in physical appearance. In order to ensure the objectivity of evaluation, the Sponsor, investigators, and other persons involved in the subject evaluation and trial implement (e.g., the Sponsor, subjects, investigators, clinical research associates, data managers, statistician, etc.) should be blinded. Blinded persons including investigators should not try to identify the group of subjects. Blind codes encrypted electronically will be stored in the Sponsor's department of medicine supply during clinical trials, and unblinding is not allowed before database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Antimicrobial Peptide PL-5 Topical Spray: 1 mg/g (1‰) (Experimental): Eligible subjects will be randomized (1:1:1) to receive twice a day, 14 days treatment of Antimicrobial Peptide PL-5 Topical Spray (1‰)
  Interventions: Drug: Antimicrobial Peptide PL-5 Topical Spray and Placebo
- Antimicrobial Peptide PL-5 Topical Spray:2 mg/g (2‰) (Experimental): Eligible subjects will be randomized (1:1:1) to receive twice a day, 14 days treatment of Antimicrobial Peptide PL-5 Topical Spray (2‰)
  Interventions: Drug: Antimicrobial Peptide PL-5 Topical Spray and Placebo
- Topical placebo (vehicle) (Placebo Comparator): Eligible subjects will be randomized (1:1:1) to receive twice a day, 14 days treatment of Antimicrobial Placebo of Antimicrobial Peptide PL-5 Topical Spray (vehicle).
  Interventions: Drug: Antimicrobial Peptide PL-5 Topical Spray and Placebo

INTERVENTIONS:
Drug: Antimicrobial Peptide PL-5 Topical Spray and Placebo — Antimicrobial Peptide PL-5 Topical Spray At about 5 cm vertically above the wound, the investigator sprays antimicrobial peptide PL-5 topical spray on the test wound. The cover area after spraying is a cone with a surface diameter of about 5 cm and area about 20 cm2. One spray dose is about 0.1 ml. The number of drug sprays is determined according to the wound area in the screening period, and the determined dose is applied consistently. During the operation, an effective spray operation is completely ejected with no leakage.
  Other Names: AMP PL-5 and Placebo

SUMMARY:
This is a Phase II, randomized, double-blind, placebo-controlled, multi-center study to evaluate the clinical efficacy and safety of Antimicrobial Peptide PL-5 Topical Spray in patients with mild infections of diabetic foot ulcers. Eligible subjects will be randomized (1:1:1) to receive twice a day, 14 days treatment of Antimicrobial Peptide PL-5 Topical Spray (1‰), Antimicrobial Peptide PL-5 Topical Spray (2‰) and topical placebo (vehicle) spray. In this study, the cut-off date for final analysis is defined as the time when all subjects have completed the last visit or discontinued the study

DETAILED DESCRIPTION:
This is a Phase II, randomized, double-blind, placebo-controlled, multi-center study to evaluate the clinical efficacy and safety of Antimicrobial Peptide PL-5 Topical Spray in patients with mild infections of diabetic foot ulcers. Approximately 90 patients (30 per treatment group) will be randomized in this study. Eligible subjects will be randomized (1:1:1) to receive twice a day, 14 days treatment of Antimicrobial Peptide PL-5 Topical Spray (1‰), Antimicrobial Peptide PL-5 Topical Spray (2‰) and placebo of Antimicrobial Peptide PL-5 Topical Spray (vehicle). In this study, the cut-off date for final analysis is defined as the time when all subjects have completed the last visit or discontinued the study. The duration of the whole study is planned for 24 months; the duration of each participant is about 4-5 weeks, including Screening period/Baseline (about 7 days), treatment period (about 14 days), Follow-up period (about 7-14 days). No interim analysis will be performed in this study. This study is a phase II study, and no statistical hypothesis is proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 65 years.
2. Non-hospitalized ambulatory subjects with Diabetes mellitus, Type I or II, according to the American Diabetes Association criteria.
3. HbA1c ≤12% at screening.
4. At baseline visit (after any required debridement), presence of Grade 2 diabetic foot infection [Grade 2 of the International Working Group on the Diabetic Foot (IWGDF) classification]

   Infection present, as defined by the presence of at least 2 of the following items:
   * Local swelling or induration
   * Erythema >0.5 cm to ≤2 cm around the ulcer.
   * Local tenderness or pain
   * Local increased warmth
   * Purulent discharge (thick, opaque to white, or sanguineous secretion)

   Mild infection of an ulcer is defined as:

   Presence of ≥2 manifestations of inflammation (purulence or erythema, tenderness, warmth, or induration), but any cellulitis/erythema extends ≤2cm around the ulcer, and infection is limited to the skin or superficial subcutaneous tissues; no other local complications or systemic illness.
5. Voluntary written consent, given before performance of any clinical investigation-related procedure not part of standard medical care, and with the understanding that consent may be withdrawn at any time without prejudice to future medical care.
6. Female subjects must meet at least one of the following additional criteria:

   * Surgically sterile with bilateral tubal ligation or hysterectomy.
   * Postmenopausal for at least one year.
   * If of childbearing potential, practicing an acceptable method of birth control for the duration of the clinical investigation as judged by the Investigator, such as condoms, foams, jellies, diaphragm, intrauterine device or abstinence

Exclusion Criteria:

1. Another cause of the inflammatory response of the skin around the ulcer (such as a trauma, gout, acute Charcot neuro-arthropathy, fracture, thrombosis, or venous stasis).
2. Foot deformities, calluses, corns, ingrown nails, fungal infections, which will impact infection or wound healing based on Investigator's judgement.
3. Received any topical or systemic antimicrobial therapy within 7 days prior to study entry (Day 1).
4. Infected diabetic foot ulcer that is associated with local wound complications such as prosthetic materials or protruding surgical hardware.
5. > 1 infected foot ulcer.
6. Concurrent or expected to require systemic antimicrobials during the study period for any infection, including diabetic foot ulcer.
7. Bone or joint involvement is suspected based on clinical examination or plain X-ray.
8. Arterial brachial index (ABI) <0.5 or ankle pressure <50 mmHg. If ABI is >1.3 (medial calcification is present), then only subjects meeting secondary testing requirements including either a toe pressure ≥30 mmHg, a transcutaneous pressure of oxygen ≥50 mmHg, or a skin perfusion pressure ≥40 mmHg are allowed. For subjects with ABI >1.3, only the initial secondary test after ABI should be used for this assessment. A documented ABI within 3 months prior to Screening is acceptable, as is the initially performed secondary testing method for subjects with ABI >1.3.
9. The subject is expected to be unable to care for the ulcer or return for all scheduled visits because of hospitalization, vacation, disability, etc. during the study period or cannot safely monitor the infection status at home.
10. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response | At EOT (End-of-therapy: within 24 hours after the final dose)
  the Investigator will grade the clinical response as （1）"infection resolved or cured" (all signs and symptoms of infection resolved);（2）"infection improving"(most, but not all, signs and symptoms of infection improved or resolved)（3）"treatment failure" (≥1 signs or symptoms of infection substantially worsening), (4)"unevaluable"(<3 days of study treatment or patient lost to follow-up), or （5）"recurrence"(a previously cured or improved infection showing worsening of signs or symptoms of infection)

SECONDARY OUTCOMES:
Microbiological response | Interim Clinical Evaluation (ICE): 7 days after the initiation of the study drug. End of Therapy (EOT): within 24 hours after the final dose. Post-therapy evaluation (PTE): 7-14 days after the final dose.
  Microbiological culture examination of wound tissue; Analysis of drug sensitivity test results; Analysis of MIC50, MIC90, geometric mean inhibitory concentration and range results of clinically isolated pathogenic bacteria. At baseline, day 1, and at all other study visits, Investigators will culture samples obtained from the wound at which culturable material and signs of infection are present. They will obtain specimens using tissue curettage with a sterile scalpel, place them into transport media, and ship them to the designated central laboratory for species identification and antibiotic susceptibility testing. For specific operations of bacteriological examination of wound tissue, please refer to the clinical microbiology operation manual. Result: 1）Resolved;2） Improved;3)Failure 4） Colonization 5） Superinfection.
Comprehensive Response | End of Therapy (EOT): within 24 hours after the final dose. Post-therapy evaluation (PTE):7-14 days after the final dose.
  At EOT and PTE, the Investigator will grade the comprehensive response as （1）"cure"(patients are clinically cured, and the bacteria are eradicated or presumed eradicated.);（2）"failure" (patients are classified as clinical failure or/and microbiological responses are failure and superinfection) or （3）"indeterminate"(if both clinical and microbiological responses are indeterminate).
Safety and tolerability | Interim Clinical Evaluation (ICE): 7 days after the initiation of the study drug. End of Therapy (EOT): within 24 hours after the final dose. Post-therapy evaluation (PTE): 7-14 days after the final dose
  The incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), and clinically significant changes in physical examination, vital signs, laboratory tests, and 12-lead electrocardiogram (ECG)
Clinical response | Interim Clinical Evaluation (ICE): 7 days after the initiation of the study drug. End of Therapy (EOT): within 24 hours after the final dose. Post-therapy evaluation (PTE): 7-14 days after the final dose.
  At each visit after enrollment, the Investigator will grade the clinical response as （1）"infection resolved or cured" (all signs and symptoms of infection resolved);（2）"infection improving"(most, but not all, signs and symptoms of infection improved or resolved)（3）"treatment failure" (≥1 signs or symptoms of infection substantially worsening), (4)"unevaluable"(<3 days of study treatment or patient lost to follow-up), or （5）"recurrence"(a previously cured or improved infection showing worsening of signs or symptoms of infection)
Wound infection Score and Total Wound Score | At baseline, day 1, and at all other study visits, investigators will compile a "total wound score" that included ratings of signs and symptoms of infection, wound measurements (maximum length, width, and depth), and assessment of granulation tissue.
  A "wound infection score" was semiquantitatively assessed by grading each of 7 parameters with a score of 0-3: (1) purulent drainage, (2) nonpurulent drainage, (3) erythema, (4) induration, (5) tenderness, (6) pain, and (7) local warmth.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - ILD Research Center, Vista, California
  - Bioresearch Partner Holdings, LLLP, Miami, Florida
  - Santos Research Center, Corp, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei Y, Li Y, Li X, Zhao Y, Xu J, Wang H, Rong X, Xiong J, Chen X, Luo G, Lv G, Lin C, Han C, Yu H, Zhang Y, Tang S, Fan Y, Tu J, Xia C, Zu H, Liu W, Liu C, Liu J, Zhang B, Nong Q, Li T, Wang L, Song G, Su Y, Chen Z, Lai W, Fu Y, Yu J, Zhang P, Yang W, Yao G, Zhang H, Fan K, Dong H, Chen Y, Wu J; PL-5 Investigators. Peceleganan Spray for the Treatment of Skin Wound Infections: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2415310. doi: 10.1001/jamanetworkopen.2024.15310. PMID 38861260
- [Background] Wei Y, Wu J, Chen Y, Fan K, Yu X, Li X, Zhao Y, Li Y, Lv G, Song G, Rong X, Lin C, Wang H, Chen X, Zhang P, Han C, Zu H, Liu W, Zhang Y, Liu C, Su Y, Zhang B, Sun B, Wang L, Lai W, Liu J, Xia C, Ji G, Zhu F, Yu J, Ahemaiti A, Dong H, Chen M; PL-5 Investigators. Efficacy and Safety of PL-5 (Peceleganan) Spray for Wound Infections: A Phase IIb Randomized Clinical Trial. Ann Surg. 2023 Jan 1;277(1):43-49. doi: 10.1097/SLA.0000000000005508. Epub 2022 Jul 4. PMID 35781462
- See also: As a library, NLM provides access to scientific literature. Inclusion in an NLM database does not imply endorsement of, or agreement with, the contents by NLM or the National Institutes of Health. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9762708/